CLINICAL TRIAL: NCT06352801
Title: Effectiveness of Self-Compassion Intervention on Enhancing Self-Compassion and Psychological Well-Being of Children With Attention Deficit/Hyperactivity Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EA230530
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: ADHD; Self-Compassion; Psychological Well-Being
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Intervention Group: In Phase 1, children participants receive a 6-session self-compassion intervention training, plus parents of the participants receive a 3-session parent group. once to twice a week, 90 minutes per session.
  Wait-list Control: receives the same intervention in Phase 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Compassion Intervention Group (Experimental): The intervention group consists of two parts: children training session and parent group sessions. All children participants will complete a total of 6 training sessions, and each session will last around 90 minutes. Parents of the children participants will also complete a total of 3 group sessions, and each session will last around 90 minutes. Participants will receive intervention in Phase 1.
  Interventions: Behavioral: Self-Compassion Intervention
- Wait-list Control Group (No Intervention): Participants will receive the same intervention in Phase 2.

INTERVENTIONS:
Behavioral: Self-Compassion Intervention — Children participants are expected to learn the concepts of self-compassion and strategies of applying self-compassion to their daily lives.
  Other Names: My DEER Compassion
  Arms: Self-Compassion Intervention Group

SUMMARY:
The study aims to investigate the underlying mechanism between Attention Deficit/Hyperactivity Disorder traits (AD/HD traits) and psychological well-being through studying the role of perceived criticism, rejection sensitivity, self-compassion and growth mindset. It also aims to explore the effectiveness of self-compassion intervention on enhancing self-compassion and psychological well-being of children with AD/HD in Hong Kong. The study will contribute to the current understanding of the supportive measures for children with AD/HD, and hopefully help to mobilize more resources to preserve children with AD/HD's mental health.

The intervention program includes the following components:

Participants will be randomly assigned to the self-compassion intervention group or the waitlist control group. The intervention group consists of two parts: children training session and parent group sessions. All children participants will complete a total of 6 training sessions, and each session will last around 90 minutes. Parents of the children participants will also complete a total of 3 group sessions, and each session will last around 90 minutes.

To investigate the intervention effectiveness, children will be asked to complete a questionnaire assessing their levels of self-compassion, emotional regulation, as well as psychological well-being in terms of life satisfaction, positive and negative affect. Parents and teachers of participants will also be asked to complete a questionnaire covering children's emotional regulation, positive and negative affect. Questionnaire data collection will be conducted prior to the intervention (i.e., Time 1), immediately after the 6-session student and 3-session parent sessions (i.e., Time 2), and 2 months after the intervention (i.e., Time 3, a 2-month follow up). It takes approximately 20-30 minutes for children and parents to complete their questionnaires.

Study Objectives:

1. To investigate the underlying mechanism of the relationship between AD/HD traits and psychological well-being
2. To explore the effectiveness of self-compassion intervention on enhancing self-compassion and psychological well-being of children with AD/HD in Hong Kong

Hypotheses:

1. AD/HD traits negatively predicts psychological well-being
2. AD/HD traits positively predicts perceived criticism or rejection sensitivity
3. Perceived criticism or rejective sensitivity negatively predicts psychological well-being
4. Perceived criticism or rejective sensitivity mediates the relationship between AD/HD traits and psychological well-being
5. Self-compassion moderates the relationship between perceived criticism or rejection sensitivity and psychological well-being
6. Growth mindset moderates the relationship between perceived criticism or rejection sensitivity and psychological well-being
7. Children with AD/HD from self-compassion intervention group yield greater improvement in self-compassion, emotional regulation and psychological well-being, than waitlist-control group.

ELIGIBILITY:
Inclusion Criteria:

* Upper primary students
* Clinical diagnosis, suspected cases of AD/HD, or having AD/HD symptoms
* Able to read, write and communicate in Chinese

Exclusion Criteria:

* Hearing, visual, or physical impairments that might hinder participation in the intervention
* Clinical diagnosis and suspected cases of Autism Spectrum Disorder (ASD)
* Prior or current participation in a psychotherapeutic treatment

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Self-Compassion Scale for Children (SCS-C) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention
  A scale consisting of 12 self-report items assessing children's self-compassion [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of self-compassion)]
Self-Compassion Scale for Children (SCS-C) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)]
  A scale consisting of 12 self-report items assessing children's self-compassion [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of self-compassion)]
Self-Compassion Scale for Children (SCS-C) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  A scale consisting of 12 self-report items assessing children's self-compassion [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of self-compassion)]
Behavioural ratings on children's executive functions | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention
  Parents and teachers will be asked to complete Behaviour Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including emotional regulation [Min. Value: 1; Max Value: 4 (with higher score indicating higher level of emotional regulation)]
Behavioural ratings on children's executive functions | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)]
  Parents and teachers will be asked to complete Behaviour Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including emotional regulation [Min. Value: 1; Max Value: 4 (with higher score indicating higher level of emotional regulation)]
Behavioural ratings on children's executive functions | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  Parents and teachers will be asked to complete Behaviour Rating Inventory of Executive Function, Second Edition (BRIEF2) measuring a range of executive functions, including emotional regulation [Min. Value: 1; Max Value: 4 (with higher score indicating higher level of emotional regulation)]
Student's Life Satisfaction Scale (SLSS) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention
  A scale consisting of 7 self-report items assessing children's life satisfaction [Min. Value: 1; Max Value: 6 (with higher score indicating higher level of life satisfaction)]
Student's Life Satisfaction Scale (SLSS) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)]
  A scale consisting of 7 self-report items assessing children's life satisfaction [Min. Value: 1; Max Value: 6 (with higher score indicating higher level of life satisfaction)]
Student's Life Satisfaction Scale (SLSS) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  A scale consisting of 7 self-report items assessing children's life satisfaction [Min. Value: 1; Max Value: 6 (with higher score indicating higher level of life satisfaction)]
Positive and Negative Affect Schedule for Children (PANAS-C/P) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention
  The PANAS, is a self-reported adjective checklist that contains two 5-item subscales designed to measure positive and negative affect. Children, parents and teachers will be asked to complete the scale [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of positive and negative affect)]
Positive and Negative Affect Schedule for Children (PANAS-C/P) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)]
  The PANAS, is a self-reported adjective checklist that contains two 5-item subscales designed to measure positive and negative affect. Children, parents and teachers will be asked to complete the scale [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of positive and negative affect)]
Positive and Negative Affect Schedule for Children (PANAS-C/P) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  The PANAS, is a self-reported adjective checklist that contains two 5-item subscales designed to measure positive and negative affect. Children, parents and teachers will be asked to complete the scale [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of positive and negative affect)]

OTHER OUTCOMES:
The Strengths and Weaknesses of Attention-Deficit/Hyperactivity Disorder Symptoms and Normal Behavior Scale (SWAN) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention
  It is an 18- question parent or teacher rating scale to assess for the indication of attention-deficit hyperactivity disorder in children [Min. Value: -3; Max Value: 3 (with lower score indicating higher level of AD/HD symptoms)]
The Strengths and Weaknesses of Attention-Deficit/Hyperactivity Disorder Symptoms and Normal Behavior Scale (SWAN) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)]
  It is an 18- question parent or teacher rating scale to assess for the indication of attention-deficit hyperactivity disorder in children [Min. Value: -3; Max Value: 3 (with lower score indicating higher level of AD/HD symptoms)]
The Strengths and Weaknesses of Attention-Deficit/Hyperactivity Disorder Symptoms and Normal Behavior Scale (SWAN) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  It is an 18- question parent or teacher rating scale to assess for the indication of attention-deficit hyperactivity disorder in children [Min. Value: -3; Max Value: 3 (with lower score indicating higher level of AD/HD symptoms)]
The Perceived Criticism Scale (PCS) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention
  The PCM is designed to provide a simple assessment of a family member's criticism from the perspective of the client/child [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of perceived criticism)]
The Perceived Criticism Scale (PCS) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)]
  The PCM is designed to provide a simple assessment of a family member's criticism from the perspective of the client/child [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of perceived criticism)]
The Perceived Criticism Scale (PCS) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  The PCM is designed to provide a simple assessment of a family member's criticism from the perspective of the client/child [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of perceived criticism)]
Children's Rejection Sensitivity Questionnaire (CRSQ) | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention
  The Children's Rejection Sensitivity Questionnaire (CRSQ) was used to assess children's rejection sensitivity in terms of anxious or angry expectations of rejection [Min. Value: 1; Max Value: 6 (with higher score indicating higher level of rejection sensitivity)]
Children's Rejection Sensitivity Questionnaire (CRSQ) | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)]
  The Children's Rejection Sensitivity Questionnaire (CRSQ) was used to assess children's rejection sensitivity in terms of anxious or angry expectations of rejection [Min. Value: 1; Max Value: 6 (with higher score indicating higher level of rejection sensitivity)]
Children's Rejection Sensitivity Questionnaire (CRSQ) | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  The Children's Rejection Sensitivity Questionnaire (CRSQ) was used to assess children's rejection sensitivity in terms of anxious or angry expectations of rejection [Min. Value: 1; Max Value: 6 (with higher score indicating higher level of rejection sensitivity)]
Growth Mindset Scale | Pre-intervention Assessment (within 4 weeks before the commencement of the intervention
  It is a 3-item Growth Mindset Scale to measure how much people believe that they can get smarter if they work at it The Children's Rejection Sensitivity Questionnaire (CRSQ) was used to assess children's rejection sensitivity in terms of anxious or angry expectations of rejection [Min. Value: 1; Max Value: 6 (with higher score indicating higher level of growth mindset)]
Growth Mindset Scale | Immediate Post-intervention Assessment (within 4 weeks after the completion of the intervention)]
  It is a 3-item Growth Mindset Scale to measure how much people believe that they can get smarter if they work at it The Children's Rejection Sensitivity Questionnaire (CRSQ) was used to assess children's rejection sensitivity in terms of anxious or angry expectations of rejection [Min. Value: 1; Max Value: 6 (with higher score indicating higher level of growth mindset)]
Growth Mindset Scale | Delayed Post-intervention Assessment (a 2-month follow up after the completion of the intervention)
  It is a 3-item Growth Mindset Scale to measure how much people believe that they can get smarter if they work at it The Children's Rejection Sensitivity Questionnaire (CRSQ) was used to assess children's rejection sensitivity in terms of anxious or angry expectations of rejection [Min. Value: 1; Max Value: 6 (with higher score indicating higher level of growth mindset)]

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Downey G, Lebolt A, Rinco´n C, Freitas AL (1998) Rejection sensitivity and children's interpersonal Dweck, C. S. (1999). Self-theories: Their Role in Motivation, Personality, and Development. Psychology Press. Ebesutani, C., Regan, J., Smith, A., Reise, S., Higa-McMillan, C., & Chorpita, B. F. (2012). The 10-item positive and negative affect schedule for children, child and parent shortened versions: application of item response theory for more efficient assessment. Journal of Psychopathology and Behavioural Assessment, 34, 191-203. Hooley, J. M., & Teasdale, J. D. (1989). Predictors of relapse in unipolar depressives: expressed emotion, marital distress, and perceived criticism. Journal of Abnormal Psychology, 98(3), 229. Huebner, E. S. (1991). Initial development of the student's life satisfaction scale. School Psychology International, 12(3), 231-240. Lai, K. Y., Leung, P. W., Luk, E. S., Wong, A. S., Law, L. S., & Ho, K. K. (2013). Validation of the Chinese strengths and weaknesses of ADHD-symptoms and normal-behaviours questionnaire in Hong Kong. Journal of Attention Disorders, 17(3), 194-202. Raes, F. (2010). Ruminating and worrying as mediators of the relationship between self-compassion and anxiety and ' depression. Personality and Individual Differences, 48, 757-761.